CLINICAL TRIAL: NCT05330416
Title: Randomized Comparison of Quality of Life With or Without Automatic Seton Placement in Perianal Crohn's Fistula
Brief Title: Comparison of Quality of Life With or Without Automatic Seton Placement in Perianal Crohn's Fistula
Acronym: SOPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOPA
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Crohn Disease
Keywords: Quality of life; Surgery; Seton
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, single-center, controlled, superiority study comparing quality of life in two groups of patients operated on for ano-perineal suppuration in Crohn's disease:
  * Flattening of the suppuration and drainage with a suture (reference strategy)
  * Flattening of the suppuration without drainage with a nipple (evaluated strategy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Reference Strategy (Active Comparator): Detailed examination of the suppuration and drainage with a seton
  Interventions: Device: Group Reference Strategy
- Group test strategy (Experimental): Detailed examination of the suppuration without drainage via a seton
  Interventions: Other: Group Test Strategy

INTERVENTIONS:
Device: Group Reference Strategy — Patients undergoing surgery for anoperineal suppuration in the context of Crohn's disease with detailed examination of the suppuration and drainage with a seton.
  Arms: Group Reference Strategy
Other: Group Test Strategy — Patients undergoing surgery for anoperineal suppuration in the context of Crohn's disease with detailed examination of the suppuration without drainage via a seton.
  Arms: Group test strategy

SUMMARY:
In patients with Crohn's disease, anal fistulas are usually treated in three stages: 1) close examination of the fistula and drainage with a seton, 2) pharmacological treatment of the inflammatory component, and 3) closure of the fistulous tract by a sphincter-sparing technique. Setons are used to ensure the permeability of the fistulous tract, to decrease the rate of re-intervention due to the formation of new abscesses or tracts. A seton is a small, often elastic, thread used for drainage. It is inserted into the fistulous tract, passing from the external orifice of the fistula (close to the anus or, in some cases, the vaginal) through the fistula and exiting via the anal orifice.

Seton use seems to minimize colonization of the mucosa of the fistulous tract by the intestinal flora, leukocyte infiltration, and the spread of inflammation within the fistulous tract. Most clinical practice guidelines advocate the use of a seton, but the level of evidence for the efficacy of this approach remains low (D, EL5). Indeed, only a few open studies have reported seton use to be potentially beneficial. In the retrospective study of 32 patients by Regueiro et al., a surgery group with seton insertion before treatment with infliximab was compared with a group on infliximab, without a seton, from the outset. Response rates were better in the group of patients with a seton, with a lower rate of recurrence and a longer time to recurrence than for the seton-less group. Another retrospective study by Schwartz et al. compared two groups - seton (n = 326) and no seton (n = 1519) - in patient with at least six months of biotherapy in three states of the USA. There were more hospitalizations and higher costs generated by greater use of the healthcare system in the group treated without a seton than in those with a seton.

The systematic use of setons in the context of Crohn's disease was inspired by the management of cryptoglandular fistula. However, the protective value of setons in this context remains far from clear, due to a lack of studies providing high-level evidence. Furthermore, the impact of seton use on patient quality of life has been little evaluated.

Investigators aim to determine whether the insertion of one or more setons in anal fistulas in Crohn's disease patients significantly alters patient quality of life. Investigators will perform a randomized controlled trial comparing two strategies: drainage surgery with and without seton use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an anal fistula requiring surgical management in the context of Crohn's disease, with or without anti-TNF treatment (infliximab or adalimumab)
* Patient over 16 years of age (for minors, the consent of one of the parents will be requested)
* Patient with health insurance coverage
* French-speaking patient
* Signed written informed consent

Exclusion Criteria:

* Patient already included in a type 1 interventional research protocol (RIPH1)
* Patient under guardianship or curatorship
* Patient incarcerated
* Patient under legal protection
* Patient refusing randomization or follow-up
* Patient refusing the medical protocol for anti-TNF treatment (infliximab or adalimumab)
* Patient already experiencing treatment failure on optimized infliximab treatment; by contrast, those experiencing treatment failure on adalimumab alone may be included
* Patient allergic or intolerant to the two anti-TNF agents (infliximab and adalimumab)
* Patient with a stoma
* Patient with an ano-recto-vaginal fistula
* Patient with anal or rectal stenosis
* Patient with ileo-anal anastomosis
* Patient without preoperative MRI

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-05-24 (Estimated); Study Completion 2025-05-24 (Estimated)

PRIMARY OUTCOMES:
Quality of life in Crohn's disease patients undergoing surgery for an anal fistula | Month 12
  This outcome corresponds to the comparison of quality of life with The Crohn's Anal Fistula Quality of Life (CAF-QoL) scale with 28 simple questions covering three areas: fistula-related symptoms, treatment-related symptoms and quality of life. The CAF-QoL scale is ready for use as a PROM in research and clinical practice. It complements objective clinical evaluation of fistula by capturing impact on the patient.

SECONDARY OUTCOMES:
Clinical cure rate at 6 months | Month 6
  This outcome corresponds to Clinical cure defined by: absence of seton, closure of secondary orifices, absence of leakage under pressure and absence of new suppuration.
Clinical cure rate at 12 months | Month 12
  This outcome corresponds to Clinical cure defined by: absence of seton, closure of secondary orifices, absence of leakage under pressure and absence of new suppuration.
Rate of re-interventions for the drainage of a new abscess or a new fistula at 12 months | Month 12
  This outcome corresponds to the Number of re-interventions for the drainage of a new abscess and/or fistula (operations to close the fistulous tract excluded).
Radiological cure rate, as determined by MRI at 12 months | Month 12
  This outcome corresponds to the absence of T2 hyperintensity, contrast uptake after injection of gadolinium and abscess > 2 cm.
Rate of use of sphincter-sparing techniques at 12 months | Month 12
  This outcome corresponds to the rate of use of sphincter-sparing techniques (simple removal of the seton, rectal lowering flap, FiLaC laser, biological glue, intersphincter ligation of the fistulous tract, injection of mesenchymal stem cells).
Clinical and radiological cure rate at 12 months in the group of patients receiving an injection of mesenchymal stem cells | Month 12
  This outcome corresponds to the Clinical and radiological cure rate (pre-defined criteria).

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Fathallah, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Torres J, Bonovas S, Doherty G, Kucharzik T, Gisbert JP, Raine T, Adamina M, Armuzzi A, Bachmann O, Bager P, Biancone L, Bokemeyer B, Bossuyt P, Burisch J, Collins P, El-Hussuna A, Ellul P, Frei-Lanter C, Furfaro F, Gingert C, Gionchetti P, Gomollon F, Gonzalez-Lorenzo M, Gordon H, Hlavaty T, Juillerat P, Katsanos K, Kopylov U, Krustins E, Lytras T, Maaser C, Magro F, Marshall JK, Myrelid P, Pellino G, Rosa I, Sabino J, Savarino E, Spinelli A, Stassen L, Uzzan M, Vavricka S, Verstockt B, Warusavitarne J, Zmora O, Fiorino G. ECCO Guidelines on Therapeutics in Crohn's Disease: Medical Treatment. J Crohns Colitis. 2020 Jan 1;14(1):4-22. doi: 10.1093/ecco-jcc/jjz180. No abstract available. PMID 31711158
- [Background] Adamina M, Bonovas S, Raine T, Spinelli A, Warusavitarne J, Armuzzi A, Bachmann O, Bager P, Biancone L, Bokemeyer B, Bossuyt P, Burisch J, Collins P, Doherty G, El-Hussuna A, Ellul P, Fiorino G, Frei-Lanter C, Furfaro F, Gingert C, Gionchetti P, Gisbert JP, Gomollon F, Gonzalez Lorenzo M, Gordon H, Hlavaty T, Juillerat P, Katsanos K, Kopylov U, Krustins E, Kucharzik T, Lytras T, Maaser C, Magro F, Marshall JK, Myrelid P, Pellino G, Rosa I, Sabino J, Savarino E, Stassen L, Torres J, Uzzan M, Vavricka S, Verstockt B, Zmora O. ECCO Guidelines on Therapeutics in Crohn's Disease: Surgical Treatment. J Crohns Colitis. 2020 Feb 10;14(2):155-168. doi: 10.1093/ecco-jcc/jjz187. PMID 31742338
- [Background] Bouchard D, Abramowitz L, Bouguen G, Brochard C, Dabadie A, de Parades V, Eleouet-Kaplan M, Fathallah N, Faucheron JL, Maggiori L, Panis Y, Pigot F, Roumeguere P, Senejoux A, Siproudhis L, Staumont G, Suduca JM, Vinson-Bonnet B, Zeitoun JD. Anoperineal lesions in Crohn's disease: French recommendations for clinical practice. Tech Coloproctol. 2017 Sep;21(9):683-691. doi: 10.1007/s10151-017-1684-y. Epub 2017 Sep 19. PMID 28929282
- [Background] Lee MJ, Heywood N, Sagar PM, Brown SR, Fearnhead NS; pCD Collaborators. Surgical management of fistulating perianal Crohn's disease: a UK survey. Colorectal Dis. 2017 Mar;19(3):266-273. doi: 10.1111/codi.13462. PMID 27423057
- [Background] Gecse KB, Bemelman W, Kamm MA, Stoker J, Khanna R, Ng SC, Panes J, van Assche G, Liu Z, Hart A, Levesque BG, D'Haens G; World Gastroenterology Organization, International Organisation for Inflammatory Bowel Diseases IOIBD, European Society of Coloproctology and Robarts Clinical Trials; World Gastroenterology Organization International Organisation for Inflammatory Bowel Diseases IOIBD European Society of Coloproctology and Robarts Clinical Trials. A global consensus on the classification, diagnosis and multidisciplinary treatment of perianal fistulising Crohn's disease. Gut. 2014 Sep;63(9):1381-92. doi: 10.1136/gutjnl-2013-306709. Epub 2014 Jun 20. PMID 24951257